CLINICAL TRIAL: NCT01066416
Title: Effects of Endoscopic Sinus Surgery for Chronic Sinusitis on Asthma Control
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Endeavor Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Asthma; Chronic Sinusitis
MeSH Terms: conditions — Asthma | interventions — Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medical therapy (Placebo Comparator): Patients undergo surgery 6 months after randomization
  Interventions: Other: medical therapy
- Surgery (Experimental): Patients undergo surgery at time of randomization
  Interventions: Procedure: Endoscopic Sinus Surgery

INTERVENTIONS:
Procedure: Endoscopic Sinus Surgery
  Arms: Surgery
Other: medical therapy — Subjects will undergo surgery 6 months after randomization
  Arms: Medical therapy

SUMMARY:
It is unknown whether surgical treatment of chronic sinusitis improves asthma control in patients with poorly controlled asthma. This is a randomized trial of surgical plus medical sinus therapy versus medical therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: General

  1. 18 years of age or older
  2. Women need one of the following: negative pregnancy test or suitable birth control or post-menopausal status
  3. Informed consent and ability to comply with study procedures
  4. Patients must meet inclusion criteria for both asthma and sinus disease.

Inclusion criteria: Asthma

In order to qualify for the 6 week run-in, patients must have poorly controlled asthma as defined by the following criteria:

1. Diagnosis of asthma confirmed either by demonstrating a positive methacholine challenge test (defined as a decrease in FEV1 by at least 20%, following administration of 8mg or less of inhaled methacholine) or a positive bronchodilator response (defined as a change from base line of >12% and at least 200ml in either FEV1 or FVC, following administration of a short-acting, inhaled bronchodilator).
2. Either:

   * Asthma Control Questionnaire score > 1.5 or
   * Use of inhaled rescue ß-agonist >/= 16 puffs per week (excluding use as a pre-medication for exercise; 1 nebulizer treatment = 2 puffs of inhaler) at any time during the past month or
   * >1 hospitalization or unscheduled MD visit in the past 6 months for asthma symptoms or
   * >1 course of oral steroid use in past 6 months or
   * > 2 weeks of systemic steroids in last 6 months.

Exclusion Criteria:

1. Current smokers or those with at least a 10 pack-year smoking history
2. Presence of any concurrent diseases that, in the investigator's opinion, would interfere with participation in the study or that might put the participant at risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Asthma Control Score

CONTACTS AND LOCATIONS:
Locations (1):
- Evanston Hospital, Evanston, Illinois, United States